CLINICAL TRIAL: NCT07289256
Title: Comparison of Hip Spica Duration (6 Weeks vs 12 Weeks) Following Open Reduction and Pelvic Osteotomy in Developmental Dysplasia of the Hip
Brief Title: Does a 6-week Duration of Hip Spica Immobilization Provide Comparable Clinical and Radiological Outcomes to 12 Weeks in Children Undergoing Open Reduction and Pelvic Osteotomy for Developmental Dysplasia of the Hip (DDH)?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Makarious Medhat Mahfouz Ishak, resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Spica cast and DDH
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: DDH

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups to receive either 6 weeks or 12 weeks of hip spica immobilization following open reduction for developmental dysplasia of the hip (DDH)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-week spica group (Experimental): Patients will undergo open reduction and pelvic osteotomy for DDH, followed by immobilization in a hip spica cast for 6 weeks.
  Interventions: Procedure: hip spica immobilization for 6 weeks
- 12-week spica group (Experimental): Patients will undergo open reduction and pelvic osteotomy for DDH, followed by immobilization in a hip spica cast for 12 weeks.
  Interventions: Procedure: hip spica immobilization for 12 weeks

INTERVENTIONS:
Procedure: hip spica immobilization for 6 weeks — Patients undergo open reduction and pelvic osteotomy for DDH followed by hip spica cast immobilization for 6 weeks.
  Arms: 6-week spica group
Procedure: hip spica immobilization for 12 weeks — Patients undergo open reduction and pelvic osteotomy for DDH followed by hip spica cast immobilization for 12 weeks.
  Arms: 12-week spica group

SUMMARY:
The study aim is to compare clinical and radiological outcomes of 6-week versus 12-week hip spica immobilization following open reduction and pelvic osteotomy for DDH.

DETAILED DESCRIPTION:
Developmental dysplasia of the hip (DDH) is a common pediatric orthopedic disorder with a prevalence of 2% to 3% in neonates. Surgical intervention, including open reduction and pelvic osteotomy, is indicated when closed reduction fails or diagnosis is delayed. Traditionally, postoperative immobilization in a hip spica cast is recommended for 12 weeks to maintain stability. However, recent studies suggest that shorter durations (6 weeks) may provide equivalent stability with fewer complications such as joint stiffness, muscle atrophy, skin breakdown, and caregiver burden. some fractures occurs after the cast, according to Alassaf 2018 out of total of 128 patients (162 hips) 93 were in the double-leg spica group, and 69 were in the single-leg spica group three patients had a greenstick distal femur fracture after double-leg spica and one after single-leg spica. There is no international consensus on the optimal spica duration, and evidence is limited. Proving that 6 weeks immobilization is not inferior to 12 weeks immobilization could improve outcomes, reduce costs, and lessen morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Children 18 months-6 years undergoing open reduction with pelvic osteotomy for DDH.

Exclusion Criteria:

* • Infection

  * Paralytic hip dislocation

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Redislocation rate | 12 months post-surgery
  Incidence of hip redislocation within the first 12 months after open reduction and hip spica immobilization.

SECONDARY OUTCOMES:
Radiological outcomes | 3, 6, and 12 months post-surgery
  Assessment of acetabular index and femoral head position using pelvic X-rays at follow-up
Functional outcomes | Within 6-12 months post-surgery
  Time to independent ambulation and hip joint range of motion assessment.
Complications | During immobilization period and up to 3 months post-cast removal
  Occurrence of cast-related problems including skin sores, pressure ulcers, and cast intolerance.